CLINICAL TRIAL: NCT05823987
Title: A Phase II Study of Oncolytic Virotherapy Combined With Tislelizumab Plus Lenvatinib in Patients With Advanced Biliary Tract Cancer
Brief Title: Oncolytic Virotherapy Combined With Tislelizumab Plus Lenvatinib in Patients With Advanced Biliary Tract Cancer (OPTIONS-05)
Acronym: OPTIONS-05
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2302270-6
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Advanced Biliary Tract Cancer
MeSH Terms: interventions — tislelizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H101 + Tislelizumab+ Lenvatinib (Experimental): H101 intratumorally injection starts at day 0. Tislelizumab plus lenvatinib will be initiated on day 1. Tislelizumab will be administered at 200 mg i.v. every 3 weeks plus a lenvatinib (bodyweight ≥ 60 kg, 12 mg; < 60 kg, 8 mg) orally daily every 3 weeks until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: H101; Drug: Tislelizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: H101 — a modified human recombinant type 5 adenovirus with genetic modifications
  Other Names: Oncorine
Drug: Tislelizumab — a PD-1 immune check inhibitor
Drug: Lenvatinib — Lenvatinib capsules

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of oncolytic virotherapy combined with Tislelizumab plus lenvatinib in patients with advanced biliary tract cancer (BTC).

DETAILED DESCRIPTION:
Recent studies have suggested that local destruction of tumor tissue by oncolytic virus induced activation and maturation of dendritic cells and tumor-specific T cells by cross-presentation of tumor antigens. While pd-1 blocking antibody interferes with PD-1 mediated T-cell regulatory signaling. And combination of pd-1 blocking antibody plus lenvatinib showed increased ORR in many type of human cancers. Therefore, the objective of this study is to evaluate the efficacy and safety of oncolytic virotherapy combined with Tislelizumab plus lenvatinib in patients with advanced BTC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry.
* Participants must have unresectable or metastatic histologically or cytologically confirmed biliary tract cancer (BTC)
* Participants must have failed 1 line of systemic regimens for advanced BTC due to disease progression or toxicity.
* At least one measurable site of disease as defined by RECIST criteria with spiral CT scan or MRI.
* Performance status (PS) ≤ 2 (ECOG scale).
* Life expectancy of at least 12 weeks.
* Adequate blood count, liver-enzymes, and renal function: absolute neutrophil count ≥ 1,500/L, platelets ≥75 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula )
* Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion Criteria:

* History of cardiac disease, including clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment
* Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
* Prior treatment with oncolytic virotherapy.
* Radiotherapy administered less than 4 weeks prior to study treatment start.
* Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
* Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
* Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to:

  1. history of interstitial lung disease
  2. Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection)
  3. known acute or chronic pancreatitis
  4. active tuberculosis
  5. any other active infection (viral, fungal or bacterial) requiring systemic therapy
  6. history of allogeneic tissue/solid organ transplant
  7. diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of Tislelizumab treatment.
  8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study.
  9. Live vaccine within 30 days prior to the first dose of Tislelizumab treatment or during study treatment.
  10. History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of Tislelizumab treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS
* Medication that is known to interfere with any of the agents applied in the trial.
* Any other efficacious cancer treatment except protocol specified treatment at study start.
* Patient has received any other investigational product within 28 days of study entry.
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by investigator.

SECONDARY OUTCOMES:
Duration of Response (DOR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DOR is defined as the time from first documented complete or partial response until disease progression, death from any cause, or censoring at date of last tumor assessment.
Progression Free Survival (PFS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  PFS is defined as the time from study treatment to disease progression or all-cause death as assessed by the investigator (whichever occurs first)
Overall survival (OS) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  OS is defined as the time from study treatment to the date of death of the subject, regardless of the cause of death
Disease control rate (DCR) evaluated by the investigator per Response Evaluation Criteria in Solid Tumors Version 1.1 | max 24 months
  DCR is defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | max 42 months
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience at least one AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, Principal Investigator — Fudan University Shanghai Cancer Center, Shanghai
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No